CLINICAL TRIAL: NCT06181773
Title: Development and Feasibility Testing of Intervention on Improving Caregivers' Perception of Preschool Child Weight and Their Feeding Practices in Yangzhou City, China
Brief Title: Empowering Parents to Optimize Feeding Practices With Preschool Children (EPO Feeding Program)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: King's College London (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 20231019
Record Dates: First submitted 2023-11-20; First posted 2023-12-26 (Actual); Last update posted 2024-08-13 (Actual); Status verified 2023-10

CONDITIONS: Feeding Practices
Keywords: Feeding practices; Preschool children; Group-based training program; Caregivers; Parents; Weight perception

STUDY DESIGN:
Intervention Model Description: The participants will be randomly allocated to two arms: the intervention group and the control group.
Who Masked: Outcomes Assessor
Masking Description: Due to the nature of the study, only the research members who collect and analyze the data from participants can be masked to the randomization.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- EPO Feeding program + Usual care (intervention group) (Experimental): Participants in the intervention group will receive the EPO Feeding program and usual care. EPO Feeding program includes four, weekly group training sessions for parents of preschool children (aged 2-6) led by healthcare professionals. The intervention incorporates lessons and information (i.e., slide shows and handouts), group discussions, motivational interviewing, and other supplementary materials (e.g., stories, key messages, and educational videos) to improve parents' knowledge, skills, and behaviors regarding feeding preschool children. After each module, homework activities will be assigned to participants to help reinforce their knowledge, skills, and behaviors. The motivational interviewing will be conducted by healthcare professionals to provide individual support. Moreover, a WeChat group will be set up to facilitate parental involvement, learning, and communication.
  Interventions: Behavioral: EPO Feeding Program
- Usual care (control group) (No Intervention): Parents involved in the control group will receive usual care, which is the printed materials of child health-related dietary recommendations published by the Chinese government/Nutrition Society. These materials will also be distributed to the participants in the intervention group. After the final data collection at one-month follow-up, participants from this control group will be offered the complete material package of the EPO Feeding program, their child's weight status measured at the final time point and provided access to pre-recorded modules by healthcare professionals as a incentive.

INTERVENTIONS:
Behavioral: EPO Feeding Program — The EPO Feeding program focused on providing parents with information based on scientific evidence and the most current nutritional recommendations regarding positive feeding practices and healthy eating during the preschool years.
  Arms: EPO Feeding program + Usual care (intervention group)

SUMMARY:
Parental feeding practices are critical in shaping preschool children's eating habits and preventing childhood obesity. However, parents frequently adopt inappropriate feeding practices that are not optimal for their children's health and may result in children's nutrition-related problems. Thus, the research team developed a psychoeducational intervention - Empowering Parents to Optimize Feeding Practices with Preschool Children (EPO Feeding program) to support healthier feeding practices. The primary objective of this study is to test the feasibility and acceptability of the EPO Feeding program. The secondary objective is to test the potential effects of the EPO Feeding program against a control group, on parental feeding practices, parental perception of their child's weight, parenting sense of competence, their child's eating behaviors, and their child's BMI-Z scores.

DETAILED DESCRIPTION:
The development process of the EPO Feeding program was conducted according to the MRC framework and included a systematic review of the relevant literature and stakeholder participation through qualitative interviews with parents and healthcare professionals and focus groups with kindergarten staff. The cross-sectional study was also conducted to determine if parental perception of child weight had a close link to their specific feeding practices. It also provided information on the frequency of specific feeding practices in the research setting, which aided inform the prioritization of intervention content. After structuring the EPO Feeding program, more stakeholders were engaged to further refine the intervention before designing the feasibility RCT.

After completing the baseline assessment, parents of preschool children who are responsible for their child's eating behaviors and family food environment will be randomized and allocated to one of the groups through a concealed computerized random number generator. Participants in the intervention group will receive the EPO Feeding program and usual care. EPO Feeding program includes four, weekly group training sessions for parents of preschool children (aged 2-6) led by healthcare professionals. The intervention incorporates lessons and information (i.e., slide shows and handouts), group discussions, motivational interviewing, and other supplementary materials (e.g., stories, key messages, and educational videos) to improve parents' knowledge, skills, and behaviors regarding feeding preschool children. After each module, homework activities will be assigned to participants to help reinforce their knowledge, skills, and behaviors. The motivational interviewing will be conducted by healthcare professionals to provide individual support. Moreover, a WeChat group will be set up to facilitate parental involvement, learning, and communication. Parents will complete the measures immediately after the 4-week program, and at one-month follow-up.

The primary outcomes are i) feasibility measured through retention rates and adherence; ii) acceptability of the program to parents and the healthcare professionals delivering the program through an anonymous survey, qualitative process evaluation, and fidelity of intervention delivery. The secondary outcomes focus on the potential program effects on i) parental feeding practices; ii) parents' accurate perception of their child's weight; iii) parenting sense of competence; iv) parental accounts of their child's eating behaviors; and v) children's BMI-Z scores.

ELIGIBILITY:
Parents Inclusion Criteria:

1. Parents who are the caregivers (caregivers (i.e., parents who are responsible for the family food environment and their preschool children's eating
2. One of their children aged 2 to 6 years (if (more than) two preschool children, the parent is instructed to focus on the child whose eating, nutrition or weight status they are more concerned about)
3. Parents are aged ≥18 years
4. Able to provide informed consent
5. Able to speak and write Chinese

Exclusion Criteria:

1. Parents with diagnosed severe mental illness such as schizophrenia, uncontrolled bipolar disorder, or mental retardation that would prevent participation in the feasibility intervention.
2. Their preschool children with diseases that influence their eating and nutrition (e.g., diagnosed eating disorders).
3. Parents who have eating disorders or are pregnant during the study period.
4. Parents or parents with children who are participating in another intervention related to child growth and nutrition.
5. Parents who have participated in previous aspects of the intervention development (e.g., focus groups).

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 84 (Actual)
Dates: Start 2023-12-08 (Actual); Primary Completion 2024-03-07 (Actual); Study Completion 2024-03-31 (Actual)

PRIMARY OUTCOMES:
Retention rate | Record in each module (week 1,2,3,4); retention rate will be caculated after completing intervention (week4)
  The percentage of participants who complete the intervention.
Attendance/Adherence | Attendance record in each module (week 1,2,3,4)
  Number of modules attended
Recruitment rate | Baseline
  Recruitment rates: The percentage of participants take part in the intervention.
Participants Acceptance of Intervention | Week 4 (after intervention)
  An anonymous survey containing eight closed questions (e.g., How would you rate the quality of the program? How valuable was the program in helping you optimise feeding practices?) and one open question (i.e., comments on the experiences or feelings about the program) after the intervention. Each item is rated on a 10-point Likert scale. The acceptability will be calculated by averaging the scores of all the items with higher scores indicating greater acceptability of the program.
Participants Acceptance of Intervention2 | Week 4,5 (after intervention)
  Process evaluation of the program: semi-structured interviews with participants. The interview topic guide will be used to instruct the interview (e.g., participants' advice and suggestions on the program, outcome measures, and randomization).
Provider Acceptance of Intervention (healthcare professionals) | Week 4,5 (after intervention)
  Process evaluation of the program: semi-structured interviews with healthcare professionals who will deliver the program (e.g., their advice and suggestions on the program).
The completion rates of the outcome measures | Baseline, after intervention (week 4), and one-month follow-up (week 8,9)
  The percentage of the participants complete the questionnaires at each time point.

SECONDARY OUTCOMES:
Parental feeding practices | Baseline, after intervention (week 4), and one-month follow-up (week 8,9)
  The Chinese Preschoolers' Caregivers' Feeding Behavior Scale (CPCFBS) will be used to evaluate parental restrictive feeding, pressure to eat, monitoring, encouragement of healthy eating and modeling. The Chinese version of the Child Feeding Questionnaire (C-CFQ) will be used to assess use of food as a reward. Each item of CPCFBS and C-CFQ is rated on a 5-point Likert scale. The response options for each item are 1"never", 2"rarely", 3"sometimes", 4"usually", and 5"always". Each subscale is calculated by averaging the scores of all the items in that subscale with higher scores indicating a greater prevalence of that feeding practice. (positive/responsive feeding: monitoring, encouragement of healthy eating and modeling; negative/non-responsive feeding: restrictive feeding, pressure to eat and reward)
Parental accurate perception of preschool child weight (self-reported) | Baseline, after intervention (week 4), and one-month follow-up (week 8,9)
  The Chinese version of the Child Feeding Questionnaire (C-CFQ) will be used to measure self-reported perception of child weight by asking, "How would you describe your child's weight?". Each item is rated on a 5-point Likert scale. The responses include 1"very underweight," 2"slightly underweight," 3"normal weight," 4"slightly overweight," and 5"very overweight."
  Parental accurate perception of child weight was assessed by determining the discrepancy between their perceptions of child weight and the child's actual weight status. A score of zero indicated non-misperceptions, while negative or positive scores indicated misperceptions.
Parental accurate perception of child weight (visual) | Baseline, after intervention (week 4), and one-month follow-up (week 8,9)
  Parental visual perception of child weight will be assessed by the perception of Healthy Weight (PPHW) in the age range 2 to 6 years old. The parent will be asked to select one gender from an appropriate image/sketch that most closely matches the child's body type on a 7-point scale (1 = a severely underweight child, 4 = an average-weight child, 7 = an obese child).
  Parental accurate perception of child weight was assessed by determining the discrepancy between their perceptions of child weight and the child's actual weight status. A score of zero indicated non-misperceptions, while negative or positive scores indicated misperceptions.
Parenting Sense of Competence | Baseline, after intervention (week 4), and one-month follow-up (week 8,9)
  The Chinese version of Parenting Sense of Competence Scale will be used to assess parental perception of their abilities to manage the demands of parenting. It includes two subscales: Efficacy and Satisfaction. Each item is rated on a 6-point Likert scale from "Absolutely disagree" to "Absolutely agree". Each subscale is calculated by averaging the scores of all the items in that subscale with higher scores indicating a greater efficacy and satisfaction of parenting role.
Child eating behaviors | Baseline, after intervention (week 4), and one-month follow-up (week 8,9)
  Five types of child eating behaviors are assessed by the Chinese Preschoolers' Eating Behavior Questionnaire (CPEBQ), including food fussiness, satiety responsiveness, food responsiveness, emotional eating and initiative eating. Each item is rated on a 5-point Likert scale with higher scores indicating a greater prevalence of that eating behavior. The response options for each item are 1"never", 2"rarely", 3"sometimes", 4"usually", and 5"always". Each subscale is calculated by averaging the scores of all the items in that subscale. (positive eating behaviors: initiative eating; negative eating behaviors: food fussiness, satiety responsiveness, food responsiveness, and emotional eating)
Child weight status | Baseline, after intervention (week 4), and one-month follow-up (week 8,9)
  BMI Z-scores are categorized into three groups: underweight (Z-score < -2), normal weight (-2 ≤ Z-score ≤ 1), overweight (1 < Z-score ≤ 2) and obese (Z-score > 2)

OTHER OUTCOMES:
The feasibility and acceptability of EPO Feeding program: Observation checklist | Week 1,2,3,4 (record in each intervention)
  Process evaluation: observation checklist. The researcher will make fieldnotes about the module delivery and responses to the modules provided on the program, barriers and enablers of the program completion, participants' task engagement and its overall structure, delivery, and content of the program.
The feasibility and acceptability of EPO Feeding program: Fidelity checklist | Week 6-7 (after intervention)
  The fidelity checklist of the EPO Feeding program delivery will be used to measure how closely they adhere to the manual and the underpinned theoretical models. All modules will be audio recorded by a facilitator and watched by another researcher to rate against the fidelity checklists and ensure modules are delivered as intended.
The feasibility and acceptability of EPO Feeding program: Progress criteria assessment | Week 13-14 (after follow-up measurement)
  Pre-specified criteria used to inform progression to a definitive RCT

CONTACTS AND LOCATIONS:
Overall Officials: Jian Wang, Principal Investigator — King's College London
Locations (1):
- YangZhou Baoying Maternal and Child Health Hospital, Yangzhou, Jiangsu, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Wang J, Chang YS, Wei X, Cao Y, Winkley K. Feasibility of a Psychoeducational Intervention for Empowering Parents to Optimise Feeding Practices in China: A Randomised Controlled Feasibility Trial. Matern Child Nutr. 2026 Mar;22(1):e70155. doi: 10.1111/mcn.70155. PMID 41503735
- [Derived] Wang J, Cao Y, Wei X, Winkley K, Chang YS. Empowering parents to optimize feeding practices with preschool children (EPO-Feeding): A study protocol for a feasibility randomized controlled trial. PLoS One. 2024 Jun 3;19(6):e0304707. doi: 10.1371/journal.pone.0304707. eCollection 2024. PMID 38829882